CLINICAL TRIAL: NCT03927612
Title: Virtual Reality to Improve Social Perspective Taking in Youth With Disruptive Behavior Disorders
Brief Title: Virtual Reality to Improve Social Perspective Taking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tom Hummer, Assistant Research Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1902596251
Record Dates: First submitted 2019-04-18; First posted 2019-04-25 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Conduct Disorder; Child; Adolescent; Attention Deficit and Disruptive Behavior Disorders; Child Behavior Disorders; Virtual Reality; Social Perception; Magnetic Resonance Imaging
Keywords: virtual reality; perspective taking; conduct disorder; oppositional defiant disorder; functional magnetic resonance imaging; child; adolescent
MeSH Terms: conditions — Conduct Disorder; Attention Deficit and Disruptive Behavior Disorders; Child Behavior Disorders; Oppositional Defiant Disorder

STUDY DESIGN:
Intervention Model Description: This project will examine how levels of a virtual reality treatment that provides users with the alternate perspective of an interpersonal interaction impacts psychological and neurobiological markers of perspective taking. Following the initial screening visit, participants will be randomly assigned to different VR perspective conditions, stratified by sex, presence/absence of ADHD diagnosis, and ODD/CD diagnosis, via an a priori randomization chart. An equal number of youth will be randomly assigned to either the alternate perspective condition or control condition. Visits 1 and 2 will be identical for both groups. At Visit 3, the initial VR scenarios and assessments will be identical. The participant will then re-experience the VR scenarios depending on their assigned condition. Additional VR assessments and the MRI scan will be identical for both groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Assignment will be sealed for the experimenter until immediately prior to Visit 3 (for visit preparation, experimenter must be unblinded).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Alternate Perspective (Experimental): After experiencing VR scenarios, participants will experience the interactions again from the virtual counterpart's perspective within the VR system.
  Interventions: Device: Virtual reality perspective taking training
- Control Perspective (Placebo Comparator): After experiencing VR scenarios, participants will experience the interactions again from the same perspective in the VR system.
  Interventions: Device: Virtual reality control perspective

INTERVENTIONS:
Device: Virtual reality perspective taking training — Virtual reality system provides first-person perspective of a virtual social interaction in a school cafeteria as the subject attempts to complete a goal. A virtual counterpart interferes with this goal. In the alternate perspective condition, participants will then experience the scenario again from the counterpart's perspective, including internal thoughts of the virtual counterpart.
  Arms: Alternate Perspective
Device: Virtual reality control perspective — Virtual reality system provides first-person perspective of a virtual social interaction in a school cafeteria as the subject attempts to complete a goal. A virtual counterpart interferes with this goal. In the control perspective condition, participants will then experience the scenario again from identical perspective.
  Arms: Control Perspective

SUMMARY:
This project will examine how virtual reality treatment that provides users with the alternate perspective of a virtual interpersonal interaction impacts psychological and neurobiological markers of social perspective taking in children with a disruptive behavior disorder. The investigators anticipate that experiencing a virtual encounter from a counterpart's point-of-view improves a child's perspective taking and alters brain function related to imagining another person's pain.

DETAILED DESCRIPTION:
Oppositional defiant disorder (ODD) and conduct disorder (CD), collectively known as disruptive behavior disorders (DBDs), involve persistent physical or verbal confrontations, antisocial behavior, and emotional outbursts. Despite a range of biological and environmental risk factors for DBD, social-cognitive impairments are a common link, and improving these deficits should be beneficial for all patients with DBD.

Children and adolescents with DBD have deficits in social perspective taking that contribute significantly to these behavior problems. Perspective taking is the ability to perceive the world from another person's point of view, including making inferences about the capabilities, feelings, and expectations of others. Perspective taking requires substantial motivation and cognitive resources and can be difficult to achieve, particularly for children. A failure to understand or value another person's perspective inhibits helping behavior without clear direct benefits. Perspective taking skills are related to empathic concern, which encompasses feelings of sympathy and concern for unfortunate others, and theory of mind, the ability to accurately infer others' mental states, such as intentions. Negative attribution biases are more likely in individuals with poor theory of mind. Thus, improving children's perspective-taking skills should allow them to better understand a counterpart's thinking and intentions, increasing empathic concern, and reducing hostile attribution biases-and therefore improving the likelihood that prosocial behavior occurs.

In the brain, perspective taking engages circuitry underlying empathic concern and theory of mind. In fMRI studies, imagining pain to the self or other, often in conjunction with images depicting painful scenarios, engages the brain's salience network. Dorsal ACC and bilateral anterior insula, the regions most commonly activated in response to other's pain, also show strong responses to self-perspective pain. However, in youth with DBD, there is a decreased response to other-perspective pain in dACC and anterior insula, despite no change or a heightened response to self-perspective pain.

Software interventions have shown some promise to improve perspective taking. In particular, VR has exciting therapeutic potential to address perspective-taking deficits because it provides naturalistic yet controlled environments in which users can experience interactions from multiple viewpoints. VR interventions typically provide better generalization to real-world behavioral changes compared to traditional methods. VR has an advantage over traditional interventions because it provides an embodied experience that is a middle ground between therapy room settings and the real world (e.g., school, home) where problematic behaviors occur.

In this investigation, the investigators will build upon a current VR design using an Oculus Quest virtual reality headset. After experiencing virtual interpersonal conflicts in a school cafeteria setting, participants will re-experience scenarios in one of two manners: an enriched perspective from the virtual counterpart's point-of-view, with internal dialogue and background information; or a control perspective, which replays the original point-of-view. During this proof-of-concept phase, the primary target is social perspective taking. The investigators will assess functional engagement of this target by quantifying (1) the ability to recognize and understand the virtual counterpart's perspective; and (2) the neural response (in pain circuitry) to pain experienced by the virtual counterpart, a common marker for perspective taking that is abnormal in DBD.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9-12
* English-speaking
* Meet DSM-5 criteria for oppositional defiant disorder (ODD), conduct disorder (CD), or Other Specified or Unspecified Disruptive, Impulse-Control, and Conduct Disorder
* Right-handed
* Estimated full-scale IQ greater than 70

Exclusion Criteria:

* Bipolar disorder, any disorder involving psychosis, pervasive developmental disorders, current or past substance use disorder, or current major depressive disorder
* History of neurological problems (e.g., epilepsy, traumatic brain injury)
* Contraindications for MRI
* Sibling who has participated in this study
* Experience negative side effects during use of virtual reality (e.g., VR sickness)
* In opinion of investigator, cannot complete study procedures or is inappropriate for study participation

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom A Hummer, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Health Neuroscience Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Families underwent clinical interview to establish child's psychiatric diagnoses (required disruptive behavior disorder without autism spectrum disorder or current depression for assignment to group). Participants also underwent baseline surveys, practice VR (also used to assess presence of VR sickness for exclusion criteria), and baseline MRI scan. Enrolled participants were not randomized if they did not meet inclusion criteria or discontinued participation prior to the intervention visit.
Period: Overall Study
Arm/Group | Alternate Perspective | Control Perspective
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: While all participants completed the study, data from one participant in the Alternate Perspective arm was not included in analysis due to inability to follow instructions and two participants in the Control Perspective were not included (one failure to follow instructions; one equipment malfunction).
Groups:
- Total: Total of all reporting groups
Arm/Group | Alternate Perspective | Control Perspective | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 22 | 45
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.87 (1.00) | 11.16 (1.03) | 11.01 (1.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 15 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 18 | 16 | 34
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-intervention on the Virtual Reality Perspective Taking Scale
Description: This scale provides a 0-100 score that indicates the degree to which participants understand the perspective of their virtual counterpart, derived from the Perspective Taking subscale of the Interpersonal Reactivity Index. A higher change score indicate greater improvement in perspective taking in the virtual environment. The scale will be completed twice on the same day, before and after the intervention.
Time Frame: 1 Day
Population: Children aged 9-12 with a disruptive behavior disorder
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Alternate Perspective | Control Perspective
Number analyzed (Participants) | 23 | 22
Score on a scale | 16.3 (27.9) | -10.4 (26.3)

2. Primary Outcome: Change From Pre-intervention on the Acknowledgement of Other Perspective Scale
Description: This scale allows participants to rate the relative importance of the virtual counterpart's perspective, on a 0-100 scale, with a scenario-specific question. A higher change score indicates greater improvement in acknowledging the virtual counterpart's perspective. The scale will be completed twice on the same day, before and after the intervention.
Time Frame: 1 Day
Population: Children aged 9-12 with a disruptive behavior disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alternate Perspective | Control Perspective
Number analyzed (Participants) | 23 | 22
score on a scale | 2.0 (27.1) | -1.4 (18.5)

3. Primary Outcome: Change From Pre-intervention in Brain Activity in Response to Self Pain vs. Other Pain
Description: Functional magnetic resonance imaging (fMRI) will measure the blood-oxygen level-dependent (BOLD) response in the dorsal anterior cingulate cortex, left anterior insula, and right anterior insula while imagining pain happening to oneself or the virtual counterpart. Perspective taking and empathy are reflected by a similar BOLD response to self and other pain. This score reflects the change from baseline in the Self Pain - Other Pain contrast in each region. A lower score to Self vs. Other pain results from a stronger response to other's pain, reflecting improved perspective taking. Therefore, lower values reflect a stronger neural response to other's pain, compared to the baseline visit.
Time Frame: The fMRI scans will be administered 0-2 weeks prior to the intervention and the day of the intervention (upon completion of the intervention).
Population: Children aged 9-12 with a disruptive behavior disorder
Measure: Mean (Standard Deviation); unit: BOLD signal change (Self vs. Other Pain)
Arm/Group | Alternate Perspective | Control Perspective
Number analyzed (Participants) | 20 | 18
BOLD signal change (Self vs. Other Pain)
  Left Anterior Insula Change | 0.089 (0.19) | -0.070 (0.25)
  Right Anterior Insula Change | 0.078 (0.22) | -0.128 (0.30)
  Dorsal Anterior Cingulate Cortex Change | 0.10 (0.27) | -0.080 (0.34)

ADVERSE EVENTS:
Time Frame: 1 Day
Description: Adverse events are only collected for events occurring post-randomization, including during and immediately after the intervention on the day of the study visit.
Arm/Group | Alternate Perspective | Control Perspective
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT03927612/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03927612/ICF_000.pdf